CLINICAL TRIAL: NCT04448366
Title: Cognitive Behavioral Therapy to Improve Quality of Life After Surgical Treatment of Women With Endometriosis
Brief Title: Cognitive Behavioral Therapy in Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: Radboud University Medical Center (Other); Catharina Ziekenhuis Eindhoven (Other); Jeroen Bosch Ziekenhuis (Other); Isala (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-1464
Record Dates: First submitted 2020-06-03; First posted 2020-06-25 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Endometriosis; Quality of Life; Pain
Keywords: Endometriosis; Cognitive behavioral therapy; Quality of life
MeSH Terms: conditions — Endometriosis; Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral therapy group (Experimental): Patients in this group will undergo a total of 7 sessions of CBT in 5 months in addition to usual care.
  Interventions: Behavioral: Cognitive behavioral therapy
- Usual care (No Intervention): Patients in this group will undergo usual care only.

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Patients in the CBT group will receive usual care. In addition, they will undergo one pre-surgery and six post-surgery face-to-face sessions of CBT. In the pre-surgery session, management of expectations towards surgery will be addressed. In the six post-surgery sessions, attention will be paid to psycho-education concerning the biological link between endometriosis-related pain and stress, relaxation training, cognitive stress management, and management of anxiety, catastrophizing and hypervigilance. The CBT sessions will be coordinated by a registered psychotherapist who is experienced in CBT and has knowledge about endometriosis. All CBT will be individual sessions.
  Arms: Cognitive behavioral therapy group

SUMMARY:
Endometriosis affects 10% of reproductive aged women and causes severe pain and impaired quality of life (QoL). Surgery for endometriosis results in long term symptom relief in only 40% of women.

QoL in endometriosis improves after surgery, but not to the level of healthy women. Mediators in QoL include pain intensity, pain cognitions, and stress. In a preliminary study, patients with negative pain cognitions reported higher pain intensities compared to patients with positive pain cognitions. This indicates that psychological factors explain considerable variance in pain, suggesting that changing these factors by psychological interventions may contribute to improving QoL. Cognitive behavioral therapy (CBT) is proven effective as a psychological treatment for pain-related symptoms. The primary objective of this study is to investigate whether usual care combined with CBT improves QoL in patients undergoing surgery for endometriosis compared to usual care only. Secondary objectives are to investigate whether pain intensity, pain cognitions, perceived stress, fatigue and objectively measured cortisol levels mediate the effects of CBT on QoL in both groups.

In a randomized controlled trial, 100 endometriosis patients undergoing surgery will be randomized between usual care with CBT (CBT group) and usual care only (control group). Women in the CBT group will receive, in addition to usual care, one pre-surgery and six post-surgery sessions of CBT, aimed at positively influencing mediators of QoL. Women in the control group will receive only usual care. Follow-up will be 7,5 months. In both groups QoL, pain intensity, pain cognitions, fatigue, perceived stress (using questionnaires) and objective stress (assessing cortisol in a hair sample) will be assessed at baseline assessment, T1 (two weeks after completion of all CBT sessions) and T2 (follow-up). Recruitment and treatment of patients will take place in Rijnstate hospital and Radboud University Medical Center (UMC).

DETAILED DESCRIPTION:
Rationale: Endometriosis affects 10% of reproductive aged women and causes severe pain and impaired quality of life (QoL). Surgery for endometriosis results in long term symptom relief in only 40% of women. QoL in endometriosis improves after surgery, but not to the level of healthy women. Mediators in QoL include pain intensity, pain cognitions, and stress. In a preliminary study, patients with negative pain cognitions reported higher pain intensities compared to patients with positive pain cognitions. This indicates that psychological factors explain considerable variance in pain, suggesting that changing these factors by psychological interventions may contribute to improving QoL. Cognitive behavioral therapy (CBT) is proven effective as a psychological treatment for pain-related symptoms. QoL after surgery for endometriosis should be improved. Pain cognitions could be psychosocial targets in the treatment of endometriosis related symptoms. We hypothesize that CBT focusing on cognitions towards pain for women undergoing surgery for endometriosis improves pain cognitions, leading to improvement of QoL.

Objective: The primary objective of this study is to investigate whether usual care combined with CBT improves QoL in patients undergoing surgery for endometriosis compared to usual care only. Secondary objectives are to investigate whether pain intensity, pain cognitions, perceived stress, fatigue and objectively measured cortisol levels mediate the effects of CBT on QoL in both groups.

Study design: In a randomized controlled trial, 100 endometriosis patients undergoing surgery will be randomized between usual care with CBT (CBT group) and usual care only (control group). Women in the CBT group will receive, in addition to usual care, one pre-surgery and six post-surgery sessions of CBT, aimed at positively influencing mediators of QoL. Women in the control group will receive only usual care. Follow-up will be 7,5 months. In both groups QoL, pain intensity, pain cognitions, fatigue, perceived stress (using questionnaires) and objective stress (assessing cortisol in a hair sample) will be assessed at baseline assessment, T1 (two weeks after completion of all CBT sessions) and T2 (follow-up). Recruitment and treatment of patients will take place in Rijnstate hospital and Radboud University Medical Center (UMC).

Study population: Healthy female volunteers aged 18-50 years with an indication for endometriosis surgery due to endometriosis associated pain.

Intervention: Cognitive behavioral therapy administered in a total of seven sessions.

Main study parameters/endpoints: The difference in Quality of Life at the last measurement compared to baseline assessment.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The control group will receive usual care. The intervention group will receive usual treatment plus a total of seven sessions of CBT. In addition, all participants are asked to fill in seven questionnaires at baseline assessment, T1 (two weeks after completion of all CBT sessions) and T2 (follow-up): the EHP-30, SF-36, PSC, PASS, CIS, NRS and PSS. Furthermore, the researcher will carefully collect a scalp hair sample of at least 0,5 cm thickness. This will be done at baseline assessment, T1 and T2. The hair sample will be analyzed for cortisol levels in a laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 50 years
* Proven endometriosis (by ultrasound, MRI or surgery)
* An indication for endometriosis debulking surgery* due to endometriosis-related pain
* Being able to understand, read and write Dutch * An indication for surgery is present when hormonal and/or analgesic therapy failed in suppressing pain symptoms.

Exclusion Criteria:

* An mood, anxiety or personality disorder diagnosis according to the DSM-5 at the moment of inclusion
* Undergoing psychological treatment at the moment of inclusion
* Use of psychopharmacologic medication aimed at altering mood at the moment of inclusion Patients that have endometriosis-related unwanted childlessness only
* Chronic pain (3 days a week for at least 6 months) that can be allocated to other diseases or syndromes
* Scalp hair shorter than 4 cm

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Change in Health Related Quality of Life assessed by the Endometriosis Health Profile 30 | 7,5 months
  The Endometriosis Health Profile 30 (EHP-30) is a disease-specific QoL questionnaire which is validated for use in endometriosis patients and measures the impact of the disease on physical, mental and social aspects of life.
  The EHP-30 is not a numerical scale.
Change in general Quality of Life assessed by the Short Form 36 | 7,5 months
  The Short Form 36 (SF-36) is a multipurpose, general health survey which is applied to measure QoL on nine different domains: physical functioning, social functioning, role limitations due to physical health, role limitations due to emotional problems, emotional well-being, vitality, pain, general health, and health change.
  The SF-36 is not a numerical scale.

SECONDARY OUTCOMES:
Change in Pain intensity assessed by the Numerical Rating Scale | 7,5 months
  The Numerical Rating Scale (NRS) ranges from 0 (no pain) to 10 (unbearable pain), and is the most commonly used subjective measure to assess pain intensity. Patients will score there estimated average pain intensity and there highest pain intensity of the previous 7 days.
  Minimum value: 0 Maximum value: 20 Higher score indicates a higher level of pain intensity.
Change in Subjective stress assessed by the Perceived Stress Scale | 7,5 months
  Perceived stress will be measured using the Perceived Stress Scale (PSS), a 10-item validated psychological instrument for measuring nonspecific perceived stress. Items are designed to score how unpredictable, uncontrollable, and overloaded respondents find their lives.
  Minimum value: 10 Maximum value: 50 Higher score indicates a higher level of perceived stress.
Change in Objective stress assessed by measuring scalp hair cortisol levels | 7,5 months
  Cortisol will be extracted from hair. The researcher will carefully collect a scalp hair sample of at least 0,5 cm thickness and sent these to the laboratory to analyze. The most proximal part represents the most recently grown piece of hair. Hair samples will be cut into a segment corresponding to the 4 cm closest to the scalp, reflecting cortisol secretion over the four months prior to sample collection. Cortisol extraction from hair will be carried out using an enzyme-linked immunoassay (ELISA).
Changes in pain cognitions assessed by the Pain anxiety symptom scale | 7,5 months
  The Pain anxiety symptom scale (PASS) measures anxiety caused by pain. Questions are asked about feelings of fear of pain, cognitive anxiety, avoidance behaviour, and physiological anxiety symptoms.
  Minimum value: 0 Maximum value: 200 Higher score indicates a higher pain anxiety.
Changes in pain cognitions assessed by the pain catastrophizing Scale | 7,5 months
  The pain catastrophizing Scale (PCS) measures the degree of pain catastrophizing of the participant by measuring elements of helplessness and pessimism in relation to the ability to cope with the pain experience.
  Minimum value: 0 Maximum value: 52 Higher score indicates a higher level of catastrophizing
Changes in Fatigue assessed by the checklist individual strength | 7,5 months
  The checklist Individual Strength (CIS) is a 20-item questionnaire addressing fatigue, concentration, motivation and activity over the past two weeks.
  The CIS is not a numerical scale.

CONTACTS AND LOCATIONS:
Overall Officials: A W Nap, MSc, PhD, Principal Investigator — Rijnstate
Locations (5):
- Netherlands (5):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Jeroen Bosch Hospital, 's-Hertogenbosch, North Brabant
  - Catharina Hospital, Eindhoven, North Brabant
  - Isala Hospital, Zwolle, Overijsel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Aken MAW, Oosterman JM, van Rijn CM, Ferdek MA, Ruigt GSF, Peeters BWMM, Braat DDM, Nap AW. Pain cognition versus pain intensity in patients with endometriosis: toward personalized treatment. Fertil Steril. 2017 Oct;108(4):679-686. doi: 10.1016/j.fertnstert.2017.07.016. Epub 2017 Sep 11. PMID 28911933
- [Background] van Aken M, Oosterman J, van Rijn T, Ferdek M, Ruigt G, Kozicz T, Braat D, Peeters A, Nap A. Hair cortisol and the relationship with chronic pain and quality of life in endometriosis patients. Psychoneuroendocrinology. 2018 Mar;89:216-222. doi: 10.1016/j.psyneuen.2018.01.001. Epub 2018 Jan 5. PMID 29414035
- [Background] Giudice LC, Kao LC. Endometriosis. Lancet. 2004 Nov 13-19;364(9447):1789-99. doi: 10.1016/S0140-6736(04)17403-5. PMID 15541453
- [Background] Soliman AM, Yang H, Du EX, Kelley C, Winkel C. The direct and indirect costs associated with endometriosis: a systematic literature review. Hum Reprod. 2016 Apr;31(4):712-22. doi: 10.1093/humrep/dev335. Epub 2016 Feb 6. PMID 26851604
- [Background] Ehde DM, Dillworth TM, Turner JA. Cognitive-behavioral therapy for individuals with chronic pain: efficacy, innovations, and directions for research. Am Psychol. 2014 Feb-Mar;69(2):153-66. doi: 10.1037/a0035747. PMID 24547801
- [Background] Faramarzi M, Pasha H, Esmailzadeh S, Kheirkhah F, Heidary S, Afshar Z. The effect of the cognitive behavioral therapy and pharmacotherapy on infertility stress: a randomized controlled trial. Int J Fertil Steril. 2013 Oct;7(3):199-206. Epub 2013 Sep 18. PMID 24520487
- [Background] Richter J, Bittner A, Petrowski K, Junge-Hoffmeister J, Bergmann S, Joraschky P, Weidner K. Effects of an early intervention on perceived stress and diurnal cortisol in pregnant women with elevated stress, anxiety, and depressive symptomatology. J Psychosom Obstet Gynaecol. 2012 Dec;33(4):162-70. doi: 10.3109/0167482X.2012.729111. Epub 2012 Oct 19. PMID 23078196
- [Background] Archer KR, Devin CJ, Vanston SW, Koyama T, Phillips SE, Mathis SL, George SZ, McGirt MJ, Spengler DM, Aaronson OS, Cheng JS, Wegener ST. Cognitive-Behavioral-Based Physical Therapy for Patients With Chronic Pain Undergoing Lumbar Spine Surgery: A Randomized Controlled Trial. J Pain. 2016 Jan;17(1):76-89. doi: 10.1016/j.jpain.2015.09.013. Epub 2015 Oct 23. PMID 26476267
- [Background] Wang L, Chang Y, Kennedy SA, Hong PJ, Chow N, Couban RJ, McCabe RE, Bieling PJ, Busse JW. Perioperative psychotherapy for persistent post-surgical pain and physical impairment: a meta-analysis of randomised trials. Br J Anaesth. 2018 Jun;120(6):1304-1314. doi: 10.1016/j.bja.2017.10.026. Epub 2018 Feb 14. PMID 29793597
- [Derived] Boersen Z, Oosterman J, Hameleers EG, Delcliseur HSMJ, Lutters C, IJssel de Schepper A, Braat D, Verhaak CM, Nap A. Determining the effectiveness of cognitive behavioural therapy in improving quality of life in patients undergoing endometriosis surgery: a study protocol for a randomised controlled trial. BMJ Open. 2021 Dec 8;11(12):e054896. doi: 10.1136/bmjopen-2021-054896. PMID 34880026